CLINICAL TRIAL: NCT05791331
Title: A Randomized Controlled Trial of Oscillatory Mechanics Versus Oxygenation-based Criteria for Surfactant Therapy
Brief Title: REspiratory MEchanics for Delivering Individualised Exogenous Surfactant
Acronym: REMEDIES
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Collaborators: Politecnico di Milano (Other)
Responsible Party: Principal Investigator, Anna Lavizzari, Principal Investigator, Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Sperimentazione 3115; Studio Numero 6379 (Other: Comitato Etico Milano Area 2)
Record Dates: First submitted 2022-12-09; First posted 2023-03-30 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Respiratory Distress Syndrome in Premature Infant
Keywords: Surfactant; Respiratory mechanics; Respiratory Oscillometry; Forced Oscillation technique; Neonatal RDS; CPAP; CPAP failure; Premature infant
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A/Control (Active Comparator): Surfactant administration following clinical assessment
  Interventions: Other: Surfactant administration following clinical assessment
- B/Intervention (Experimental): Surfactant administration following both lung mechanics assessment and clinical assessment
  Interventions: Other: Surfactant administration following lung mechanics assessment in addition to clinical assessment

INTERVENTIONS:
Other: Surfactant administration following lung mechanics assessment in addition to clinical assessment — Surfactant is administered following oxygenation-based criteria and if the Xrs is ≤ -23.3 cmH2O*s /L
  Arms: B/Intervention
Other: Surfactant administration following clinical assessment — Surfactant is administered following oxygenation-based criteria
  Arms: A/Control

SUMMARY:
This study is an interventional, non-pharmacological, multicentric, randomized, controlled, superiority, non-profit study. Its primary objective is to evaluate if the administration of surfactant based on FOT assessment will allow a 5-day reduction in the duration of respiratory support as compared to standard practice in preterm infants between 27+0 and 32+6 weeks' gestation. The secondary objectives are:

1. to determine if a lung mechanics-based approach for administering surfactant will change treatment timing; and
2. to assess the impact of the novel approach on other neonatal general outcomes. The study will take place within the neonatal intensive care units. Non-invasive respiratory support will be delivered by nasal CPAP with a starting pressure of 5-8 cmH2O. FiO2 will be titrated in order to achieve the target SpO2 91-95%.

Infants matching the clinical criteria for inclusion will be randomized in two arms following the current data protection and confidentiality regulations. Central, computer-generated randomization (allocation 1:1) with variable block sizes according to gestational age will be used. Infants will be stratified according to gestational age (27+0 -28+6 weeks; 29+0 -30+6 weeks; 31+0 -32+6 weeks) and center.

Study Arms:

A) Surfactant administration following oxygenation-based criteria (clinical assessment) (control) B) Surfactant administration following both lung mechanics assessment OR oxygenation-based criteria (clinical assessment) (intervention).

ELIGIBILITY:
Inclusion Criteria:

1. Gestational age (GA) ≥ 27+0 and < 33+0 weeks
2. Spontaneously breathing infants, requiring non-invasive respiratory support (nasal CPAP or bilevel nasal CPAP). Criteria for commencement of non-invasive respiratory support: FiO2 >0.30 for target SpO2 88-93% or Silverman score ≥ 5.
3. Inborn
4. Written parental consent obtained
5. Administration of Caffeine bolus 20 mg/kg IV or PO as per standard care

Exclusion Criteria:

1. Major congenital anomalies
2. Need of intubation in delivery suite according to the AAP guidelines for neonatal resuscitation or early at the admission in NICU (within one hour from birth).
3. Surfactant therapy prior to the study entry
4. Severe birth asphyxia, defined by APGAR score ≤ 5 at 10 minutes after birth OR continued need for resuscitation 10 minutes after birth OR pH < 7.0 or base excess (BE) < -12 mmol/l on umbilical cord or on an arterial or capillary blood sample obtained within 1 hour from birth OR moderate to severe encephalopathy
5. Respiratory failure secondary to conditions other that RDS as identified by lung imaging (air leaks, lung malformations…)
6. Any clinical condition which may place the infants at undue risk as deemed by clinicians
7. Participation to trials with competitive outcomes or likely to have an impact on the primary outcome of the study
8. Outborn patients

Ages: 27 Weeks to 33 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 458 (Estimated)
Dates: Start 2023-05-18 (Estimated); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Days of respiratory support | From date of randomization until the date of discharge from hospital or date of death from any cause, whichever came first, assessed up to 48 months"
  Number of days of required respiratory support

SECONDARY OUTCOMES:
First surfactant administration | From date of randomization until the date of discharge from hospital or date of death from any cause, whichever came first, assessed up to 48 months"
  Time of first surfactant administration (in hours)
Days of non-invasive respiratory support | From date of randomization until the date of discharge from hospital or date of death from any cause, whichever came first, assessed up to 48 months"
  Number of days of non-invasive respiratory support
Days of invasive respiratory support | From date of randomization until the date of discharge from hospital or date of death from any cause, whichever came first, assessed up to 48 months"
  Number of days of invasive respiratory support
Patients intubated and mechanically ventilated | From date of randomization until the date of discharge from hospital or date of death from any cause, whichever came first, assessed up to 48 months"
  Number of patients intubated and mechanically ventilated
Patients receiving multiple surfactant doses | From date of randomization until the date of discharge from hospital or date of death from any cause, whichever came first, assessed up to 48 months"
  Number of patients receiving multiple surfactant doses
Days on supplemental oxygen | From date of randomization until the date of discharge from hospital or date of death from any cause, whichever came first, assessed up to 48 months"
  Number of days on supplemental oxygen
Total cumulative oxygen exposure | From date of randomization until the date of discharge from hospital or date of death from any cause, whichever came first, assessed up to 48 months"
  Total cumulative oxygen exposure computed as the time integral of the FiO2 values
Infants receiving more than 28 days of respiratory support | From date of randomization until the date of discharge from hospital or date of death from any cause, whichever came first, assessed up to 48 months"
  Number of infants receiving more than 28 days of respiratory support
Infants developing BPD | From date of randomization until the date of discharge from hospital or date of death from any cause, whichever came first, assessed up to 48 months"
  Number of infants developing BPD according to the definition by NICHD 2016
Infants developing air-leaks | From date of randomization until the date of discharge from hospital or date of death from any cause, whichever came first, assessed up to 48 months"
  Number of infants developing air-leaks
Infants developing prematurity-associated complications | From date of randomization until the date of discharge from hospital or date of death from any cause, whichever came first, assessed up to 48 months"
  Number of infants developing prematurity-associated complications (severe intraventricular haemorrhage (IVH), periventricular leukomalacia (PVL), necrotizing enterocolitis (NEC), sepsis, retinopathy of prematurity (ROP), patent ductus arteriosus requiring pharmacological or surgical treatment)
Infants discharged home with oxygen or respiratory support | From date of randomization until the date of discharge from hospital or date of death from any cause, whichever came first, assessed up to 48 months"
  Number of infants discharged home with oxygen or respiratory support
Days to achieve full-enteral feeding | From date of randomization until the date of discharge from hospital or date of death from any cause, whichever came first, assessed up to 48 months"
  Number of days to achieve full-enteral feeding (160 ml/kg/day of milk intake)
Days of hospitalization | From date of randomization until the date of discharge from hospital or date of death from any cause, whichever came first, assessed up to 48 months"
  Number of days of hospitalization
Infants receiving postnatal steroids | From date of randomization until the date of discharge from hospital or date of death from any cause, whichever came first, assessed up to 48 months"
  Number of infants receiving postnatal steroids